CLINICAL TRIAL: NCT00003002
Title: A Phase I Study of a HER-2/Neu Peptide Based Vaccine With GM-CSF as an Adjuvant in Patients With Advanced Stage HER-2/Neu Expressing Cancers
Brief Title: HER-2/Neu Vaccine Plus GM-CSF in Treating Patients With Stage III or Stage IV Breast, Ovarian, or Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14798; UW-100.1; NCI-V97-1259
Record Dates: First submitted 1999-11-01; First posted 2004-07-30 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer; Lung Cancer; Ovarian Cancer
Keywords: stage III breast cancer; stage IV breast cancer; stage III non-small cell lung cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Adenocarcinoma of Lung | interventions — sargramostim

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines made from the HER2/neu antigen may make the body build an immune response and kill tumor cells. Colony-stimulating factors such as GM-CSF increase the number of immune cells found in bone marrow or peripheral blood.

PURPOSE: Phase I trial to study the effectiveness of HER-2/neu vaccine plus GM-CSF in treating patients who have stage III or stage IV breast cancer, stage III or stage IV ovarian cancer, or stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of serial intradermal vaccinations of HER-2/neu derived peptides with sargramostim (GM-CSF) as an adjuvant in patients with stage III or IV HER-2/neu expressing breast, ovarian, or nonsmall cell lung cancer. II. Determine whether immunity can be elicited with peptides derived from the intracellular domain of the HER-2/neu protein. III. Determine whether immunity can be elicited with peptides derived from the extracellular domain of the HER-2/neu protein. IV. Determine whether cytotoxic T cells specific for the HER-2/neu protein can be elicited in patients with HLA-A2 by immunization with peptides derived from the HER-2/neu protein.

OUTLINE: Patients receive one of three HER-2/neu peptide vaccine formulations that also contain sargramostim (GM-CSF) as the vaccine adjuvant. Each vaccine is studied in 20 patients. A maximum of 3 patients receive a vaccine each month for 6 months to monitor the potential toxicity associated with sequential immunizations. Patients receive a follow-up evaluation 1 month after the last vaccination. Those patients who have an immune response related to the vaccine will continue to have immunologic evaluations performed every 2 months while immune responses can still be detected.

PROJECTED ACCRUAL: 60 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III or IV breast, ovarian, or nonsmall cell lung cancer (NSCLC): Adenocarcinoma No progressive disease May have comlpeted at least 1 standard chemotherapy regimen Confirmed HER-2/neu protein overexpression in tumor (either primary tumor or metastasis)

PATIENT CHARACTERISTICS: Age: Pre or postmenopausal Performance status: Not specified Life expectancy: At least 12 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Renal: Creatinine less than 1.5 mg/dL Creatinine clearance greater than 60 mL/min Other: No anergy (positive delayed type hypersensitivity response required to two or more common recall antigens) Female patients must be nonfertile Male patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 1 month since cytotoxic chemotherapy Endocrine therapy: At least 1 month since corticosteroid therapy Concurrent hormone therapy allowed Radiotherapy: Concurrent radiation therapy for local control of disease allowed (except as initial therapy for NSCLC) Surgery: Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1996-04; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary (Nora) L. Disis, MD, Study Chair — University of Washington
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States